CLINICAL TRIAL: NCT02222896
Title: Assessment of the Antimicrobial Efficacy of 2% CHG Cloth Preoperative Skin Preparation
Brief Title: Preoperative Chlorhexidine Gluconate (CHG) Cloth on Healthy Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medline Industries (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R13-053
Record Dates: First submitted 2014-08-10; First posted 2014-08-22 (Estimated); Results first posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2016-11

CONDITIONS: Surgery
Keywords: Preoperative surgical skin preparation
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Chlorhexidine Gluconate Cloth (Experimental): 2% CHG, single application
  Interventions: Drug: Chlorhexidine Gluconate
- Vehicle Cloth (Placebo Comparator): Excipients on cloth
  Interventions: Other: Vehicle
- Active Chlorhexidine gluconate solution (Active Comparator): Dynahex 2% CHG
  Interventions: Drug: DynaHex-2

INTERVENTIONS:
Drug: Chlorhexidine Gluconate — 2% CHG solution on cloth
  Other Names: CHG
  Arms: Chlorhexidine Gluconate Cloth
Other: Vehicle — Excipients of CHG product only
  Other Names: Control
  Arms: Vehicle Cloth
Drug: DynaHex-2 — 2% CHG solution
  Other Names: CHG 2%
  Arms: Active Chlorhexidine gluconate solution

SUMMARY:
Evaluate the effects of Chlorhexidine Gluconate (CHG) cloth on the reduction of bacteria on the skin.

DETAILED DESCRIPTION:
Examine the antimicrobial cloth effects on normal flora bacteria of the abdomen and groin areas post CHG application.

ELIGIBILITY:
Inclusion Criteria:

* Males or Females
* 16 years of age or older
* Signed informed consent
* Good Health
* Six inches of abdomen and groin areas without tattoos, or skin disorders

Exclusion Criteria:

* Dermatological Conditions
* Sensitivity to latex
* Sensitivity to CHG

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 347 (Actual)
Dates: Start 2014-08; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H Bashir, Principal Investigator — MBT
Locations (1):
- MBT, Sterling, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Data to be shared with FDA

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Upon achieving sufficient microbial growth prior to product application on either the abdomen, groin or both abdomen and groin regions, sites of the participant were then randomized to receive one or two products for evaluation for up 4 sites. Differences in the number of participants is based on microbial qualification.
Pre-assignment Details: The sites of the participant were tested for microbial activity after product application. In some instances, more than one product could have been applied to a participant but only one product per site (groin and/or abdomen sites). Up to 4 sites could be treated: 1)both groin and abdomen, 2) only the groin or 3) only the abdomen.
Units Other Than Participants: Sites
Groups:
- CHG Cloth: CHG 3 min application
- Vehicle: Vehicle, 3 min application
- Comparator CHG: CHG Comparator, 3 min application
Period: Abdomen
Arm/Group | CHG Cloth | Vehicle | Comparator CHG
Started | 253; 253 Sites | 48; 48 Sites | 253; 253 Sites
Completed (completed number is lower as some participants did not qualify for treatment day baseline) | 219; 219 Sites | 38; 38 Sites | 221; 221 Sites
Not Completed | 34; 34 Sites | 10; 10 Sites | 32; 32 Sites
Not completed — Did not qualify | 34 | 10 | 32
Period: Groin
Arm/Group | CHG Cloth | Vehicle | Comparator CHG
Started | 254; 254 Sites | 48; 48 Sites | 250; 250 Sites
Completed (completed number is lower as some participants did not qualify for treatment day baseline) | 211; 211 Sites | 39; 39 Sites | 210; 210 Sites
Not Completed | 43; 43 Sites | 9; 9 Sites | 40; 40 Sites
Not completed — Did not qualify | 43 | 9 | 40

BASELINE CHARACTERISTICS:
Groups:
- CHG, Vehicle, Comparator CHG: Single applications of products. 3 min application for CHG and Vehicle. Comparator CHG applied according to instructions.
Arm/Group | CHG, Vehicle, Comparator CHG
Number analyzed (Participants) | 347
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 317
  >=65 years | 18
Age, Continuous [Mean (Full Range); unit: years] | 35 [16 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138
  Male | 209
Region of Enrollment [Number; unit: participants]
  United States | 347

OUTCOME MEASURES:

1. Primary Outcome: Percent Responder Rates (%) of Bacterial Reduction on the Abdomen and Groin
Description: Percent of abdomen and groin sites that showed response (achieve a 2-Log and 3-Log reduction) respectively of bacterial flora from baseline.
  Note: the number of participants in each treatment group (abdomen and/or groin) can vary depending on whether participants achieved qualifying microbial levels.
Time Frame: 10 minutes, 6 hours, 8 hours
Population: Participants received product on up to 2 abdomen and 2 groin sites, 2 abdomen only sites or 2 groin sites only.
Measure: Number; unit: Percent of Sites
Units Other Than Participants: Sites
Groups:
- CHG Cloth Abdomen: CHG 3 min application to abdomen
- CHG Cloth Groin: CHG 3 min application to groin
- Vehicle Abdomen: Vehicle 3 min application to abdomen
- Vehicle Groin: Vehicle 3 min application to groin
- Comparator CHG Abdomen: CHG comparator applied to abdomen
- Comparator CHG Groin: CHG comparator applied to groin
Arm/Group | CHG Cloth Abdomen | CHG Cloth Groin | Vehicle Abdomen | Vehicle Groin | Comparator CHG Abdomen | Comparator CHG Groin
Number analyzed (Participants) | 253 | 254 | 48 | 48 | 253 | 250
Number analyzed (Sites) | 253 | 254 | 48 | 48 | 253 | 250
Percent of Sites
  10 min | 93 | 86 | 50 | 25 | 85 | 65
  6 hours | 100 | 100 | 98 | 100 | 100 | 100
  8 hours | 100 | 100 | 98 | 100 | 100 | 100

ADVERSE EVENTS:
Description: The total number of participants that received each product. Some participants could have received up to 2 products at the same time.
Groups:
- CHG Cloth; Vehicle; Comparative CHG: Single application
Arm/Group | CHG Cloth | Vehicle | Comparative CHG
Serious Adverse Events (participants affected / at risk) | 0/297 | 0/59 | 0/292
Other Adverse Events (participants affected / at risk) | 0/297 | 0/59 | 0/292

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Confidential information based on contract.